CLINICAL TRIAL: NCT06022653
Title: Evaluation of Patients Underwent Revascularization of Aorta or Peripheral Artery at the Peripheral Vascular Disease Center, Asan Medical Center; A Single Center, Retrospective/Prospective Observational Study.
Brief Title: Asan Aorta and Peripheral Registry
Acronym: PTA
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Seung-Whan Lee, M.D., Ph.D., Principal investigator, Asan Medical Center
Other Study IDs: 2023-1234
Record Dates: First submitted 2023-08-17; First posted 2023-09-05 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Aorta Disease; Peripheral Artery Disease
Keywords: Revascularization of Aorta or Peripheral artery
MeSH Terms: conditions — Aortic Diseases; Peripheral Arterial Disease | interventions — Therapeutics; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment — EVAR,TEVAR,PTA
  Other Names: Intervention

SUMMARY:
The purpose of this study is to evaluate the clinical results of patients who received revascularization of the aorta and peripheral artery at Asan Medical Center.

DETAILED DESCRIPTION:
This study is a single center retrospective and prospective observational study to evaluate the clinical results of patients who received revascularization of the aorta and peripheral artery at asan medical center.

Data will be collected on approximately 6,000 subjects in asan medical center. Individuals will be followed up at 1, 6, and 12 months, 3, 5years up to 10 years by telephone call or hospital visit.

Data collected during all follow-up visits will include a composite of major adverse limb events, or death from any cause.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent Revascularization of Aorta or Peripheral artery from 2011 at the Peripheral Vascular Disease Center, Asan Medical Center
* Patients with aortic and peripheral artery disease are defined as:

Thoacic aorta disease/ abdominal aorta disease

1. Aneurysm
2. Aortic dissection
3. Penetrating aortic ulcer

Peripheral artery occlusive disease

1. Chronic Limb-Threatening Ischemia
2. Claudication
3. Acute limb ischemia

Exclusion Criteria:

* For prospective cohort, not agreeing to participate with written informed consent form

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent Revascularization of Aorta or Peripheral artery from 2011 at the Peripheral Vascular Disease Center, Asan Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2034-12-30 (Estimated); Study Completion 2044-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of death from any cause | 10years
  all-cause death
Rate of major Adverse Limb Events | 10years
  above-ankle amputation of the index limb,major index-limb reintervention including new bypass,interposition graft revision,thrombectomy, or thrombolysis

SECONDARY OUTCOMES:
Rate of death from all cause including cardiovascular death | 10years
  cardiovascular death,Non-cardiovascular death
Rate of stroke | 10years
  Ischemic , hemorrhagic , mixed Stroke
Rate of myocardial Infarction | 10years
  Spontaneous MI
Rate of vascular complication | 10years
  Vascular complication
Rate of bleeding | 10years
  TIMI bleeding
Success of the procedure | 10years
  PTA (target artery path) TEVAR and EVAR if aneurysm is diagnosed (the endograft is deployed accurately and the aneurysm is excluded from the circulation), if dissection is diagnosed(closure of the primary entry tear (i.e. absence of type Ia endoleak) and induction of false lumen thrombosis)
Rate of limb amputation | 10years
  Additional limb amputation of the index limb,Additional limb amputation of the non-index limb
Rate of reintervention of aorta , reintervention of index limb or non-index limb | 10years
  Reintervention of aorta , reintervention of index limb or non-index limb

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Whan Lee, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided